CLINICAL TRIAL: NCT06910423
Title: Comparative Effectiveness of the Mahayana Buddhist Awareness Training Program and Qigong Intervention on the Psychological and Neurological Outcomes for People With Insomnia: A Randomized Controlled Trial
Brief Title: Buddhist Awareness Training Program and Qigong Psychosocial Interventions for People With Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Professional and Continuing Education Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC_ETH_H_274
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Insomnia; Randomised Controlled Trial
Keywords: Mahayana Buddhist Awareness Training Program; Electroencephalography; Qigong; Hong Kong
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mahayana Buddhist Awareness Training Program (ATP) (Experimental): The 8-session ATP intervention consists of six 3-hour workshops plus two full day retreats. It will be delivered by instructors, who are trained by ATP co-founders. Participants will be guided to cultivate wisdom of non-attachment and compassion progressively by learning, contemplation, and practice. They will learn and memorize a core Buddhist mantra "Om mani padme hum," attend lectures, practice meditation, participate in experiential and reflective learning activities, and join the group discussions. Each workshop will typically begin with a sharing session followed by a Q&A segment to address participants' questions and concerns. To deepen their learning experience, revision exercises and corrections to revision exercises will be embedded at the end of each workshop. Participants will also receive guided meditation audio tracks, handouts, and weekly homework assignment to support their practice outside of workshop sessions.
  Interventions: Behavioral: Psychosocial intervention
- Qigong Intervention (Experimental): The 8-session Qigong intervention, with reference to the Five Elements Balance Qigong, will be delivered by instructors, who are trained by an experienced Daoist Qigong master teacher. It consists of six-3 hour workshops plus two full day retreats. Each workshop will typically begin with an introduction to some basic Traditional Chinese Medicine and Qigong concepts, or precautions in doing Qigong exercises and addressing participants' inquiries. Participants will progressively learn ten forms of simple Qigong movements that aim to enhance the flow of qi .The participants will also be asked to practice Qigong at home for 30 minutes at least three times per week and complete a practice log. Participants will also receive handouts to support their learning after each session.
  Interventions: Behavioral: Psychosocial intervention

INTERVENTIONS:
Behavioral: Psychosocial intervention — Culturally relevant psychosocial intervention for people with insomnia

SUMMARY:
This study aims to compare the efficacy of the Mahayana Buddhist Awareness Training Program (ATP) with a Qigong group in treating people with insomnia in Hong Kong. It also aims to investigate the underlying mechanisms, including changes in brain activity and heart rate variability during wakefulness, through which these two Eastern mind body interventions improve sleep quality. It is expected that ATP will be as efficacious as Qigong in enhancing sleep quality. Compared to the Qigong intervention, the more mind-based ATP will lead to more improvement in mental health and greater reductions in hyperarousal brain activity. Compared to ATP, the more body-based Qigong will lead to greater improvement in physical health and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* (1) being a resident of Hong Kong;
* (2) age between 50 and 75 years old;
* (3) possessing the ability to read and write in Chinese;
* (4) obtaining a Pittsburgh Sleep Quality Index (PSQI) score > 5 at baseline
* (5) demonstrating willingness to provide informed consent and adherence to study protocol.

Exclusion Criteria:

* (1) Beck Depression Inventory-II suicidal ideation score >= 2;
* (2) current use of hypnotic medications or any prescription medications that may influence sleep;
* (3) necessity to take such medications during the trial period;
* (4) ongoing therapies or clinical trials for insomnia;
* (5) intention to undergo such clinical interventions during the trial period;
* (6) working in shifts;
* (7) engagement in considerable mindfulness practices exceeding 15 minutes per day;
* (8) regular participation in different forms of Qigong, aerobics, yoga, Tai Chi, or martial arts practice at least once a week in the past six months;
* (9) limited mobility or health conditions that hinder the performance of specific Qigong movements;
* (10) currently receiving psychological, psychiatric or counselling services at least once a month;
* (11) having been diagnosed with schizophrenia or psychosis by a clinician;
* (12) having an active metal implant, pacemaker, or defibrillator in the body that affects objective assessment;
* (13) impaired skin integrity or allergies to electrode gel or adhesive at the wearable EEG device placement site;
* (14) pregnancy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes over the measurement points in the 19-item Pittsburgh Sleep Quality Index | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures sleep quality and disturbances experienced within a 1-month time frame. Scores range from 0 to 21, where a higher score represents poorer sleep quality.
Changes over the measurement points in the brain activity during wakefulness | Baseline, immediately after the intervention, 7 weeks after the intervention
  Spectral power analysis for participants' theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and gamma (30-50 Hz) bands during a 10-minute resting state wakefulness will be measured by the UMindSleep device (http://www.eegsmart.com/en/UMindSleep.html).
Changes over the measurement points in the heart rate variability | Baseline, immediately after the intervention, 7 weeks after the intervention
  This will be measured by the same wearable UMindSleep device.

SECONDARY OUTCOMES:
Changes over the measurement points in the 7-item Insomnia Severity Index | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures the nature, severity and impact of insomnia. Scores range from 0 to 28, where a higher score represents greater insomnia severity.
Changes over the measurement points in the 16-item Pre-Sleep Arousal Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures the symptoms of cognitive and somatic arousal experienced at bedtime. Scores range from 18 to 80, where a higher score represents greater pre-sleep arousal.
Changes over the measurement points in the 5-item item Santa Clara Brief Compassion Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' perceived compassion towards others. Scores ranges from 5 to 35, where a higher score represents greater compassion towards others.
Changes over the measurement points in the PROMIS® 2-item Global Physical Health-2 Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' perceived physical health. The raw total score will be converted to a T-score. T scores range from 23.4 to 63.3, where a higher score represents a higher perceived physical health.
Changes over the measurement points in the PROMIS® 2-item Global Mental Health-2 Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' perceived mental health. The raw total score will be converted to a T-score. T Scores ranges from 25.8 to 64.6, where a higher score represents a higher perceived mental health.
Changes over the measurement points in the 6-item Qi Stagnation Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' self-reported pathological qi status characterized by the slow and idle flow of qi. Scores range from 6 to 30, where a higher score represents greater qi stagnation.
Changes over the measurement points in the 6-item Qi Deficiency Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' self-reported pathological qi status characterized by the lack of qi in one of the viscera or the whole body. Scores range from 6 to 30, where a higher score represents greater qi deficiency.
Changes over the measurement points in the 2-item Generalized Anxiety Disorder-2 Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' anxiety level. Scores range from 0 to 6, where a higher score represents higher anxiety level.
Changes over the measurement points in the 2-item Patient Health Questionnaire-2 Scale | Baseline, immediately after the intervention, 7 weeks after the intervention
  It measures participants' depression level. Scores range from 0 to 6, where a higher score represents higher depression level.

OTHER OUTCOMES:
Demographics | Baseline
  Single items will be used to measure participants' age, education level, marital status, occupation, gender, presence of chronic illness, presence of life-threatening illness, and perceived energy levels throughout the day.
Treatment Acceptance | Immediately after the intervention
  This will be measured by two self-constructed items, namely, perceived helpfulness of the intervention and perceived appropriateness of the intervention content, on a 5-point Likert scale. Scores range from 2 to 10, where a higher score represents a higher treatment acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ka-Ying Dr. HUI, PhD, Principal Investigator — College of Professional and Continuing Education Limited
Locations (1):
- Division of Social Sciences, Humanities and Design, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu BWY, Gao J, Leung HK, Sik HH. A randomized controlled trial of Awareness Training Program (ATP), a group based Mahayana Buddhist intervention. Mindfulness. 2019;10:1280 1293. https://doi.org/10.1007/s12671-018-1082-1
- [Background] Ng SM, Yin MXC, Chan JSM, Chan CHY, Fong TCT, Li A, So KF, Yuen LP, Chen JP, Chung KF, Chan CLW. Impact of mind-body intervention on proinflammatory cytokines interleukin 6 and 1beta: A three-arm randomized controlled trial for persons with sleep disturbance and depression. Brain Behav Immun. 2022 Jan;99:166-176. doi: 10.1016/j.bbi.2021.09.022. Epub 2021 Oct 8. PMID 34634445
- [Background] Lee KCG, Gao J, Leung HK, Wu BWY, Roberts A, Thach TQ, Sik HH. Modulating Consciousness through Awareness Training Program and Its Impacts on Psychological Stress and Age-Related Gamma Waves. Brain Sci. 2024 Jan 17;14(1):91. doi: 10.3390/brainsci14010091. PMID 38248306
- [Background] Gao J, Leung HK, Fan J, Wu BWY, Sik HH. The neurophysiology of the intervention strategies of Awareness Training Program on emotion regulation. Front Psychol. 2022 Jul 22;13:891656. doi: 10.3389/fpsyg.2022.891656. eCollection 2022. PMID 35936346
- [Background] Chan JS, Ho RT, Wang CW, Yuen LP, Sham JS, Chan CL. Effects of qigong exercise on fatigue, anxiety, and depressive symptoms of patients with chronic fatigue syndrome-like illness: a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:485341. doi: 10.1155/2013/485341. Epub 2013 Jul 31. PMID 23983785
- [Background] Chan CS, Wong CYF, Yu BYM, Hui VKY, Ho FYY, Cuijpers P. Treating depression with a smartphone-delivered self-help cognitive behavioral therapy for insomnia: a parallel-group randomized controlled trial. Psychol Med. 2023 Apr;53(5):1799-1813. doi: 10.1017/S0033291721003421. Epub 2021 Aug 23. PMID 37310329